CLINICAL TRIAL: NCT03870880
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Intramuscular Injections of Risperidone ISM® in Patients With Acute Exacerbation of Schizophrenia: Open Label Extension (PRISMA-3_OLE)
Brief Title: Study to Evaluate the Efficacy and Safety of Risperidone ISM® in Patients With Acute Schizophrenia: Open Label Extension
Acronym: PRISMA-3_OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROV-RISP-2016-01_OLE
Record Dates: First submitted 2019-02-26; First posted 2019-03-12 (Actual); Results first posted 2022-02-23 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Masking Description: It is an open label extension
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Risperidone ISM 75 mg (Experimental): Patients assigned to this arm will receive 75 mg of Risperidone ISM during the open label extensión (OLE).
  Patients enter the study as rollover patients from the study NCT03160521, along with newly enrolled de novo patients.
  Interventions: Drug: Risperidone ISM 75 mg
- Risperidone ISM 100 mg (Experimental): Patients assigned to this arm will receive 100 mg of Risperidone ISM during the open label extensión (OLE).
  Patients enter the study as rollover patients from the study NCT03160521, along with newly enrolled de novo patients.
  Interventions: Drug: Risperidone ISM 100 mg

INTERVENTIONS:
Drug: Risperidone ISM 75 mg — Monthly (once every 4 weeks) intramuscular (IM) injection in the gluteal or deltoid muscle.
  Arms: Risperidone ISM 75 mg
Drug: Risperidone ISM 100 mg — Monthly (once every 4 weeks) IM injection in the gluteal or deltoid muscle.
  Arms: Risperidone ISM 100 mg

SUMMARY:
This is the long-term open label extension (OLE) of the study PRISMA-3 (NCT03160521). Those patients who complete participation in the main segment of the study (double blind) together with other clinically stable not previously enrolled (de novo patients) may opt to participate in this extension segment, where they will receive active Risperidone ISM® (75 mg or 100 mg)under open-label conditions every four weeks for approximately 12 months.

DETAILED DESCRIPTION:
Patients who have completed planned participation in the double-blind segment of the study PRISMA-3 (NCT03160521) through to the end of the treatment period, may be eligible to enter into this optional long-term extension segment of the study. During this extension, open-label Risperidone ISM® (i.e., either 75 or 100 mg) will be administered to all participating patients once every 4 weeks for approximately 12 months. Patients who enter into the extension segment of the study will begin participation in the extension segment immediately upon completion of the end-of-treatment visit assessments and procedures.

In addition to patients continuing from the double-blind segment of the study PRISMA-3 (rollover patients), clinically stable patients not previously enrolled in the study (de novo patients) may be eligible to enter the long-term extension segment of the study. These patients will be evaluated for eligibility at a screening visit and, if eligible, will be allocated to receive either 75 or 100 mg Risperidone ISM every 4 weeks for approximately 12 months.

Approximately 100 de novo patients are planned to be enrolled in the extension segment of the study, in addition to rollover patients.

ELIGIBILITY:
Participation in the open-label extension segment of the study PRISMA-3 is optional, and patients who complete participation in the main segment of the study (double blind segment of PRISMA-3, NCT03160521) may opt to not participate. Patients who are interested in participating must meet all eligibility criteria in order to enter into the extension segment.

Inclusion Criteria (Rollover patients):

To be eligible for entry into the extension segment of the study PRISMA-3, a patient must meet all of the following criteria at the extension baseline time point (immediately upon completion of the end-of-treatment visit assessments and procedures for the main part of the study):

1. Has completed scheduled participation in the double blind segment of the study PRISMA-3, through to the end of the treatment period and including the end-of-treatment visit
2. Continues to require long-term treatment with an antipsychotic medication, in the opinion of the investigator
3. Continues to meet contraceptive requirements of the study PRISMA-3
4. Is willing to participate in the extension segment of the study and remains capable of providing informed consent

   a. A signed informed consent form must be provided before any study assessments are performed for the extension segment
5. Continues to reside in a stable living situation, in the opinion of the investigator
6. Continues to have an identified reliable informant, in the opinion of the investigator

Exclusion Criteria (Rollover patients):

An individual who meets any of the following criteria at the extension baseline time point (immediately upon completion of the end-of-treatment visit assessments and procedures for the double blind segment PRISMA-3) will not be permitted to enter into this extension segment of the study PRISMA-3:

1. Missed more than 1 scheduled study visit during participation in the double blind segment of study PRISMA-3
2. Had an abnormal clinical laboratory value, vital sign, or ECG finding during participation in the main part of the study that, in the opinion of the investigator, was clinically relevant, related to study drug, and would compromise the well-being of the patient in the extension segment
3. Had a clinically significant or unstable medical illness/condition/disorder during the main part of the study that would be anticipated, in the investigator's opinion, to potentially compromise patient safety in the extension segment
4. Is taking or is anticipated to require any prohibited concomitant medication
5. Pregnant, lactating, or breastfeeding
6. Any contraindication for continued IM injections (e.g., treatment with anticoagulant)
7. Inadequate gluteal or deltoid musculature or excessive fat, as determined by the investigator, that would interfere with IM study drug injections
8. Study site personnel and/or persons employed by the investigator or study site or is an immediate family member of such persons

Inclusion Criteria (De Novo Patients):

1. Capable of providing informed consent
2. Age ≥ 18 and ≤ 65 years old
3. On a stable dose of oral risperidone from 4 to 6 mg daily as maintenance therapy for at least the last 4 weeks prior/before screening/baseline and would potentially benefit from conversion to an extended release injectable, in the opinion of the investigator
4. Current diagnosis of schizophrenia, according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria that is clinically stable as evidenced by:

   * No hospitalizations for acute exacerbations of schizophrenia and psychiatrically stable without significant symptom exacerbation over the last 3 months before screening based on the investigator's judgment
   * PANSS total score < 70 at screening
   * CGI-S score of ≤ 3 (mild) at screening
5. Has previously had a clinically significant beneficial response (improvement in schizophrenia symptoms), as determined by the investigator, to treatment with an antipsychotic medication other than clozapine
6. At least 2 years elapsed since initial onset of active-phase schizophrenia symptoms
7. Subject is outpatient; not hospitalized for worsening of schizophrenia within the last 3 months (hospitalization for social management within this time period is acceptable)
8. Medically stable over the last month prior to screening based on the investigator's judgment
9. BMI of 18.5 to 40.0 kg/m2 (inclusive) at screening
10. Agrees to discontinue prohibited medications as applicable and as clinically indicated according to investigator instructions
11. Dosages of all permitted medications are considered to have been stable (with the exception of medication to be used on an as-needed basis) for ≥ 2 weeks prior to the baseline visit and to remain stable during participation in this study
12. Resides in a stable living situation, in the opinion of the investigator
13. Has an identified reliable informant, in the opinion of the investigator
14. Meets the contraceptive criteria stablished in the study
15. Agrees not to post any personal medical data related to the study or information related to the study on any website or social media site during the study duration.

Exclusion Criteria (De Novo Patients):

1. History of proven inadequate clinical response to treatment with therapeutic doses (with good compliance) of risperidone or paliperidone
2. History of treatment resistance, defined as failure to respond to 2 discrete adequate trials (≥ 4 weeks with an adequate dose) of 2 different antipsychotic medications; history of clozapine use (exception: use was not because of treatment resistance or refractory psychotic symptoms)
3. Known or suspected intolerance of or allergy or hypersensitivity to risperidone, paliperidone, or any of the excipients in the IM formulations of these
4. History of neuroleptic malignant syndrome, clinically significant tardive dyskinesia or tardive dystonia
5. History of any other medical condition that is considered to pose any unjustifiable risk or interfere with study assessments
6. Clinically significant extrapyramidal symptoms at screening or baseline
7. At significant risk of suicidal, homicidal or violent ideation or behavior, by history or as clinically assessed by the investigator at screening visit
8. Answer of "yes" on item 4 or on item 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) (ideation) with the most recent episode occurring within the past 2 months, or answer "yes" to any of the 5 items (behavior) with an episode occurring within the last year
9. Current diagnosis or a history of substance use disorder according to DSM-5 criteria within 6 months prior to the screening visit (with the exception of tobacco, mild cannabis, or mild alcohol use disorder) or a positive drug screen test (with the exception of cannabis) verified by repeat testing
10. Lifetime history of diagnosis of schizoaffective disorder or bipolar disorder
11. Clinically significant comorbid neuropsychiatric disorders
12. Clinically significant or unstable medical illness/condition/disorder that would be anticipated, in the investigator's opinion, to potentially compromise patient safety or adversely affect the evaluation of efficacy
13. Laboratory abnormality that, in the opinion of the investigator, would compromise the well-being of the patient, or any of the following laboratory abnormalities at screening or baseline
14. Pregnant, lactating, or breastfeeding
15. Inadequate gluteal or deltoid musculature or excessive fat, as determined by the investigator, that would interfere with IM study drug injections
16. Any contraindication for IM injections
17. Receipt of any long-acting antipsychotic medication by IM injection within 60 days before screening
18. Current involuntary hospitalization or incarceration
19. Hospitalized for more than 30 days during the 90 days before screening
20. Participation in another clinical study in which the patient received an experimental or investigational drug or agent within 6 months before screening
21. Participation in a clinical study with Risperidone ISM within 12 months before screening
22. Study site personnel and/or persons employed by the investigator or study site or is an immediate family member of such persons
23. Patients taking or anticipated to require any prohibited concomitant medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Litman, Principal Investigator — CBH Health LLC; Yuriy Filts, Principal Investigator — CI Lviv Regional Clinical Psychiatric Hospital. Department 25
Locations (24):
- United States (13):
  - Woodland Research Northwest, Rogers, Arkansas
  - Collaborative Neuroscience Network, LLC., Garden Grove, California
  - Apostle Clinical Trials Inc., Long Beach, California
  - NRC Research Institute, Orange, California
  - CNRI-Los Angeles LLC, Pico Rivera, California
  - CNRI-San Diego, San Diego, California
  - Galiz Research, Hialeah, Florida
  - Innovative Clinical Research Inc., Hollywood, Florida
  - CBH Health LLC, Gaithersburg, Maryland
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Midwest Clinical Research Center, Dayton, Ohio
  - InSite Clinical Research, DeSoto, Texas
- Ukraine (11):
  - Regional Clinical Hospital n.a I.I. Mechnicov, Dnipro
  - Kharkiv Regional Clinical Psychiatric Hospital, Kharkiv
  - Public Healthcare Institution "Kharkiv Regional Clinical Psychiatric Hospital No. 3", Center of Urgent Psychiatry, Kharkiv
  - Kherson Regional Psychiatric Hospital, Kherson
  - Kiev City Psychiatric Hospital No. 2, Kiev
  - Kyiv Regional Medical Association "Psykhiatriya" in Kyiv, Kiev
  - CI Lviv Regional Clinical Psychiatric Hospital. Department 20, Lviv
  - CI Lviv Regional Clinical Psychiatric Hospital. Department 25, Lviv
  - Odesa Regional Medical Centre of Mental Health, Odesa
  - Maltsev Regional Clinical Psychiatric Ho, Poltava
  - N.I. Pyrogov Vinnytsya Natl Medical University, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Filts Y, Litman RE, Martinez J, Anta L, Naber D, Correll CU. Long-term efficacy and safety of once-monthly Risperidone ISM(R) in the treatment of schizophrenia: Results from a 12-month open-label extension study. Schizophr Res. 2022 Jan;239:83-91. doi: 10.1016/j.schres.2021.11.030. Epub 2021 Nov 27. PMID 34847501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enter the study as rollover patients from the previous double-blind (DB) study (NCT03160521), along with newly enrolled de novo patients. Rollover patients received Risperidone ISM in the OLE study at the same dose as during the DB study (75 mg or 100 mg). Patients who received placebo in the DB were assigned to receive either Risperidone ISM 75 or 100 mg during the OLE. De novo patients received either Risperidone ISM 75 or 100 mg depending on the previous oral risperidone treatment.
Groups:
- Rollover Placebo/Risperidone ISM 75 mg: Patients assigned to this arm were those who had been receiving placebo in the previous double-blind study and they were randomly assigned to receive Risperidone ISM 75 mg during the OLE study.
- Rollover Risperidone ISM 75mg/Risperidone ISM 75mg: Patients assigned to this arm were those who had been receiving 75 mg of Risperidone ISM in the previous double-blind study and they were randomly assigned to receive Risperidone ISM 75 mg during the OLE study.
- De Novo/Risperidone ISM 75mg: Patients assigned to this arm were de novo participants who received 75 mg of Risperidone ISM during the OLE study. Their previous oral risperidone dose was 4 mg/day.
- Rollover Placebo/Risperidone ISM 100 mg: Patients assigned to this arm were those who had been receiving placebo in the previous double-blind study and they were randomly assigned to receive Risperidone ISM 100 mg during the OLE study.
- Rollover Risperidone ISM 100 mg/Risperidone ISM 100 mg: Patients assigned to this arm were those who had been receiving 100 mg of Risperidone ISM in the previous double-blind study and they were randomly assigned to receive Risperidone ISM 100 mg during the OLE study.
- De Novo/Risperidone ISM 100 mg: Patients assigned to this arm were de novo participants who received 100 mg of Risperidone ISM in the OLE study. Their previous oral risperidone was more than 4 mg/day to a maximum of 6 mg/day.
Period: Overall Study
Arm/Group | Rollover Placebo/Risperidone ISM 75 mg | Rollover Risperidone ISM 75mg/Risperidone ISM 75mg | De Novo/Risperidone ISM 75mg | Rollover Placebo/Risperidone ISM 100 mg | Rollover Risperidone ISM 100 mg/Risperidone ISM 100 mg | De Novo/Risperidone ISM 100 mg
Started | 27 | 58 | 31 | 28 | 61 | 10
Completed | 21 | 43 | 26 | 20 | 44 | 7
Not Completed | 6 | 15 | 5 | 8 | 17 | 3

BASELINE CHARACTERISTICS:
Population: All analyses were undertaken on the population of patients who received at least one dose of study drug during the OLE study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rollover Placebo/Risperidone ISM 75 mg | Rollover Risperidone ISM 75mg/Risperidone ISM 75mg | De Novo/Risperidone ISM 75mg | Rollover Placebo/Risperidone ISM 100 mg | Rollover Risperidone ISM 100 mg/Risperidone ISM 100 mg | De Novo/Risperidone ISM 100 mg | Total
Number analyzed (Participants) | 27 | 58 | 31 | 28 | 61 | 10 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (9.29) | 40.9 (11.98) | 37.0 (10.91) | 38.4 (10.42) | 40.3 (11.04) | 35.5 (6.40) | 39.3 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 20 | 11 | 17 | 23 | 6 | 84
  Male | 20 | 38 | 20 | 11 | 38 | 4 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 0 | 2 | 0 | 0 | 8
  Not Hispanic or Latino | 26 | 53 | 31 | 26 | 61 | 10 | 207
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 0 | 6 | 14 | 0 | 32
  White | 22 | 50 | 31 | 22 | 47 | 10 | 182
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 11 | 0 | 6 | 16 | 0 | 40
  Ukraine | 20 | 47 | 31 | 22 | 45 | 10 | 175
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 27.53 (4.488) | 26.52 (4.741) | 25.28 (3.695) | 27.65 (4.954) | 27.53 (5.055) | 26.06 (3.937) | 26.88 (4.685)
Years since Schizophrenia Diagnosis [Mean (Standard Deviation); unit: years] | 11.8 (6.81) | 12.1 (9.17) | 9.6 (8.12) | 9.3 (7.45) | 11.5 (7.98) | 6.4 (5.34) | 10.9 (8.09)
Time since Acute Exacerbation or relapse (weeks) [Mean (Standard Deviation); unit: Weeks] — This is a descriptive data to show there are no differences between the treatment groups and that they are balanced at baseline.
  The acute schizophrenia was defined by:
  * Positive and Negative Syndrome Scale (PANSS) results meets:
    * Total score between 80 and 120, inclusive
    * Score of ≥ 4 (moderate or greater) for ≥ 2 of the following Positive Scale items: Item 1 (P1: delusions); Item 2 (P2: conceptual disorganization); Item 3 (P3: hallucinatory behavior); Item 6 (P6: suspiciousness/persecution)
  * Clinical Global Impression - Severity (CGI-S) score of ≥ 4 (moderately ill or worse)
  Weeks | 0.4 (0.18) | 0.3 (0.21) | 0 (0) | 0.4 (0.20) | 0.4 (0.24) | 0 (0) | 0.4 (0.21)

OUTCOME MEASURES:

1. Primary Outcome: PANSS Total Score Mean Change From Baseline to Endpoint
Description: The Positive and Negative Syndrome Scale (PANSS) is a 30-item clinician-rated instrument for assessing the symptoms of schizophrenia.The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score is the sum of all 30 PANSS items and ranges from 30 to 210, with 30 indicating absence of symptoms of schizophrenia and 210 indicating extreme ratings of all 30 symptoms. Negative change from baseline scores indicates improvements in symptoms whereas higher scores mean a worse outcome.
  Endpoint is defined as study day 365 or the last post-baseline assessment if early discontinuation.
Time Frame: Baseline and Day 365 (or the last post-baseline assessment)
Population: The analysis was undertaken on the population of patients who received at least one dose of study drug during the OLE study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Rollover Risperidone ISM 75mg/Risperidone ISM 75mg: Patients assigned to this arm were those who had been receiving 75 mg of Risperidone ISM in the previous double-blind study were randomly assigned to receive Risperidone ISM 75 mg during the OLE study.
- Rollover Placebo/Risperidone ISM 100 mg: Patients assigned to this arm were those who had been receiving placebo in the previous double-blind study and they were randomly assigned to receive either Risperidone ISM 100 mg during the OLE study.
- De Novo/Risperidone ISM 100 mg: Patients assigned to this arm were de novo participants who received 100 mg of Risperidone ISM® in the OLE study. Their previous oral risperidon was more than 4 mg/day to a maximum of 6 mg/day
Arm/Group | Rollover Placebo/Risperidone ISM 75 mg | Rollover Risperidone ISM 75mg/Risperidone ISM 75mg | De Novo/Risperidone ISM 75mg | Rollover Placebo/Risperidone ISM 100 mg | Rollover Risperidone ISM 100 mg/Risperidone ISM 100 mg | De Novo/Risperidone ISM 100 mg
Number analyzed (Participants) | 27 | 58 | 31 | 28 | 61 | 10
units on a scale | -22.9 (14.15) | -11.0 (14.52) | -0.8 (9.39) | -18.9 (14.61) | -8.7 (13.29) | -4.8 (4.80)

2. Other Pre Specified Outcome: PANSS Positive Subscale Mean Change From Baseline to Endpoint
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. In positive subscale, the 7 positive symptom constructs were: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility.
  PANSS Positive Subscale Score ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
  Endpoint is defined as study day 365 or the last post-baseline assessment if early discontinuation.
Time Frame: Baseline and Day 365 (or the last post-baseline assessment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Rollover Risperidone 75 mg/Risperidone 75 mg: Patients assigned to this arm were those who had been receiving 75 mg of Risperidone ISM in the previous double-blind study and they were randomly assigned to receive Risperidone ISM 75 mg during the OLE study.
- De Novo/Risperidone ISM 75 mg: Patients assigned to this arm were de novo participants who received 75 mg of Risperidone ISM during the OLE study. Their previous oral risperidone dose was 4 mg/day.
Arm/Group | Rollover Placebo/Risperidone ISM 75 mg | Rollover Risperidone 75 mg/Risperidone 75 mg | De Novo/Risperidone ISM 75 mg | Rollover Placebo/Risperidone ISM 100 mg | Rollover Risperidone ISM 100 mg/Risperidone ISM 100 mg | De Novo/Risperidone ISM 100 mg
Number analyzed (Participants) | 27 | 58 | 31 | 28 | 61 | 10
units on a scale | -6.0 (4.84) | -3.3 (5.47) | -0.6 (3.32) | -6.5 (5.32) | -2.6 (4.75) | -1.6 (2.67)

3. Other Pre Specified Outcome: PANSS Negative Subscale Mean Change From Baseline to Endpoint
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicated- absence of symptoms and a score of 7 indicated- extremely severe symptoms. The PANSS negative subscale score was the sum of the rating scores for the 7 negative scale items from the PANSS panel. The 7 negative symptom constructs were: blunted affect, emotional withdrawal, poor rapport, passive apathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation and stereotyped thinking. PANSS Negative Subscale Score ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
  Endpoint is defined as study day 365 or the last post-baseline assessment if early discontinuation.
Time Frame: Baseline and Day 365 (or the last post-baseline assessment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Risperidone ISM 75 mg/Risperidone ISM 75 mg: Patients assigned to this arm were those who had been receiving 75 mg of Risperidone ISM in the previous double-blind study and they were randomly assigned to receive Risperidone ISM 75 mg during the OLE study.
- Risperidone ISM 100/Risperidone ISM 100: Patients assigned to this arm were those who had been receiving 100 mg of Risperidone ISM in the previous double-blind study and they were randomly assigned to receive Risperidone ISM 100 mg during the OLE study.
Arm/Group | Rollover Placebo/Risperidone ISM 75 mg | Risperidone ISM 75 mg/Risperidone ISM 75 mg | De Novo/Risperidone ISM 75 mg | Rollover Placebo/Risperidone ISM 100 mg | Risperidone ISM 100/Risperidone ISM 100 | De Novo/Risperidone ISM 100 mg
Number analyzed (Participants) | 27 | 58 | 31 | 28 | 61 | 10
units on a scale | -4.6 (5.24) | -2.2 (3.61) | -0.3 (3.21) | -2.9 (3.75) | -2.1 (3.66) | -0.7 (4.22)

4. Other Pre Specified Outcome: PANSS General Psychopathology Subscale Mean Change From Baseline to Endpoint
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. The general psychopathology scale consists of 16 items which measure somatic concern, anxiety, guilt feelings, tension, mannerisms and posturing, depression, motor retardation, uncooperativeness, unusual thought content, disorientation, poor attention, lack of judgment and insight, disturbance of volition, poor impulse control, preoccupation and active social avoidance. PANSS General Psychopathology Subscale Score ranges from 16 (absence of symptoms) to 112 (extremely severe symptoms).
  Endpoint is defined as study day 356 or the last post-baseline assessment if early discontinuation.
Time Frame: Baseline and Day 365 (or the last post-baseline assessment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Placebo/Risperidone ISM 75 mg | Rollover Risperidone ISM 75mg/Risperidone ISM 75mg | De Novo/Risperidone ISM 75mg | Rollover Placebo/Risperidone ISM 100 mg | Rollover Risperidone ISM 100 mg/Risperidone ISM 100 mg | De Novo/Risperidone ISM 100 mg
Number analyzed (Participants) | 27 | 58 | 31 | 28 | 61 | 10
units on a scale | -12.4 (8.33) | -5.4 (7.35) | 0.2 (5.73) | -9.4 (7.43) | -3.9 (7.37) | -2.5 (2.88)

5. Other Pre Specified Outcome: Clinician Global Impression - Severity (CGI-S) Total Score Mean Change From Baseline to Endpoint
Description: The Clinician Global Impression - Severity (CGI-S) score is a 7-point clinician-rated scale for assessing the global severity of the illness. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Negative change from baseline scores indicate improvement in the severity of illness whereas higher scores mean a worse outcome.
  Endpoint is defined as study day 365 or the last post-baseline assessment if early discontinuation.
Time Frame: Baseline and Day 365 (or the last post-baseline assessment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Placebo/Risperidone ISM 75 mg | Rollover Risperidone ISM 75mg/Risperidone ISM 75mg | De Novo/Risperidone ISM 75mg | Rollover Placebo/Risperidone ISM 100 mg | Rollover Risperidone ISM 100 mg/Risperidone ISM 100 mg | De Novo/Risperidone ISM 100 mg
Number analyzed (Participants) | 27 | 58 | 31 | 28 | 61 | 10
units on a scale | -1.3 (1.02) | -0.5 (0.94) | 0.0 (0.53) | -1.0 (0.88) | -0.3 (0.80) | -0.1 (0.32)

6. Other Pre Specified Outcome: Clinician Global Impression - Improvement (CGI-I) Score
Description: The Clinical Global Impression - Improvement (CGI-I) is a single 7-point rating score total improvement, regardless of whether or not the change it is due entirely to drug treatment. Raters select one response based on the following question, "Compared to your patient's condition at the beginning of treatment, how much has your patient changed?" Scores are: 1, Very much improved; 2, Much improved; 3, Minimally improved; 4, No change; 5, Minimally worse; 6, Much worse; or 7, Very much worse.
  Endpoint is defined as study day 365 or the last post-baseline assessment if early discontinuation.
Time Frame: Day 365 (or the last post-baseline assessment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rollover Placebo/Risperidone ISM 75 mg | Rollover Risperidone ISM 75mg/Risperidone ISM 75mg | De Novo/Risperidone ISM 75mg | Rollover Placebo/Risperidone ISM 100 mg | Rollover Risperidone ISM 100 mg/Risperidone ISM 100 mg | De Novo/Risperidone ISM 100 mg
Number analyzed (Participants) | 27 | 58 | 31 | 28 | 61 | 10
score on a scale | 2.3 (1.18) | 2.9 (1.14) | 3.7 (1.09) | 2.4 (0.92) | 2.9 (1.24) | 3.1 (1.10)

7. Other Pre Specified Outcome: Overall Response Rate at Endpoint
Description: Overall response was defined as either PANSS total score ≥ 30% decrease from baseline, or CGI-I score of 2 (much improved) or 1 (very much improved).
  Endpoint is defined as study day 365 or the last post-baseline assessment if early discontinuation.
Time Frame: Day 365 (or the last post-baseline assessment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rollover Placebo/Risperidone ISM 75 mg | Rollover Risperidone ISM 75mg/Risperidone ISM 75mg | De Novo/Risperidone ISM 75mg | Rollover Placebo/Risperidone ISM 100 mg | Rollover Risperidone ISM 100 mg/Risperidone ISM 100 mg | De Novo/Risperidone ISM 100 mg
Number analyzed (Participants) | 27 | 58 | 31 | 28 | 61 | 10
percentage of participants | 74.1 [53.7 to 88.9] | 44.8 [31.7 to 58.5] | 9.7 [2.0 to 25.8] | 64.3 [44.1 to 81.4] | 45.9 [33.1 to 59.2] | 20.0 [2.5 to 55.6]

8. Other Pre Specified Outcome: Relapse Rate
Description: Relapse was defined as either increase from baseline in PANSS total score ≥30% or rehospitalization for psychotic symptoms or use of adjunctive antipsychotic medication after stabilization.
Time Frame: Day 365 (or the last post-baseline assessment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rollover Placebo/Risperidone ISM 75 mg | Rollover Risperidone ISM 75mg/Risperidone ISM 75mg | De Novo/Risperidone ISM 75mg | Rollover Placebo/Risperidone ISM 100 mg | Rollover Risperidone ISM 100 mg/Risperidone ISM 100 mg | De Novo/Risperidone ISM 100 mg
Number analyzed (Participants) | 27 | 58 | 31 | 28 | 61 | 10
percentage of participants | 11.1 [2.4 to 29.2] | 10.3 [3.9 to 21.2] | 12.9 [3.6 to 29.8] | 0 [0 to 0] | 13.1 [5.8 to 24.2] | 20.0 [2.5 to 55.6]

9. Other Pre Specified Outcome: Patients With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) is any symptom, physical sign, syndrome, or disease that either emerges during the study (from the informed consent form signature) or, if present at screening, worsens during the study, regardless of the suspected cause of the event.
  The treatment-emergent AEs (TEAEs) are defined as events that are newly occurring or worsening from the time of the first dose of the intramuscular study drug.
Time Frame: Up to Day 365 (or the last post-baseline assessment)
Population: The analysis was undertaken on the population of patients who received at least one dose of study drug during the OLE study.
  Safety data were pooled in two comparison groups (Risperidone ISM 75 mg and Risperidone ISM 100 mg) because the sample size increased and therefore the precision around the estimates.
Measure: Count of Participants; unit: Participants
Groups:
- Risperidone ISM 75 mg: Patients assigned to this arm received 75 mg of Risperidone ISM during the open label extension.
  Risperidone ISM 75 mg: Monthly (once every 4 weeks) intramuscular (IM) injection in the gluteal or deltoid muscle.
- Risperidone ISM 100 mg: Patients assigned to this arm received 100 mg of Risperidone ISM during the open label extension.
  Risperidone ISM 100 mg: Monthly (once every 4 weeks) IM injection in the gluteal or deltoid muscle.
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg
Number analyzed (Participants) | 116 | 99
Participants
  Patients with at least one TEAE | 81 | 59
  Patients with at least one treatment-related TEAE | 43 | 41
  Patients with at least one serious TEAE | 6 | 5
  Patients with at least one TEAE leading to treatment discontinuation | 7 | 8
  Patients with at least one TEAE leading to death | 1 | 0

10. Other Pre Specified Outcome: TEAEs Leading to Study Drug Discontinuation
Description: TEAEs which resulted in permanent study drug discontinuation
Time Frame: Up to Day 365 (or the last post-baseline assessment)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg
Number analyzed (Participants) | 116 | 99
Participants
  Akathisia | 0 | 1
  Diabetes mellitus | 1 | 0
  Extrapyramidal disorder | 1 | 0
  Gynaecomastia | 0 | 1
  Hepatic Steatosis | 0 | 1
  Hepatocellular injury | 0 | 1
  Libido decreased | 1 | 0
  Schizophrenia | 2 | 5
  Suicidal ideation | 1 | 0
  Weight increased | 1 | 0

11. Other Pre Specified Outcome: Patients With Treatment-related TEAEs
Description: An Adverse event (AE) is any symptom, physical sign, syndrome, or disease that either emerges during the study (from the informed consent form signature) or, if present at screening, worsens during the study, regardless of the suspected cause of the event.
  The treatment-emergent AEs (TEAEs) are defined as events that are newly occurring or worsening from the time of the first dose of the intramuscular study drug.
  The temporal relationship of the AE with the investigational medicinal product makes causality possible, and the AE cannot be due to another cause such as other drugs, a surgical intervention, or an underlying disease
Time Frame: Up to Day 365 (or the last post-baseline assessment)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg
Number analyzed (Participants) | 116 | 99
Participants
  Akathisia | 4 | 4
  Asthenia | 7 | 4
  Dizziness | 3 | 3
  Headache | 16 | 10
  Hyperprolactinemia | 11 | 10
  Insomnia | 6 | 3
  Weight increased | 6 | 3

ADVERSE EVENTS:
Time Frame: Day 1 to week 52
Groups:
- Risperidone ISM 75 mg: Patients assigned to this arm will received 75 mg of Risperidone ISM during the open label extension.
  Risperidone ISM 75 mg: Monthly intramuscular (IM) injection in the gluteal or deltoid muscle.
  Safety data were pooled in two comparison groups (Risperidone ISM 75 mg and Risperidone ISM 100 mg) because the sample size increased and therefore the precision around the estimates.
- Risperidone ISM 100 mg: Patients assigned to this arm will received 100 mg of Risperidone ISM during the open label extension.
  Risperidone ISM 100 mg: Monthly IM injection in the gluteal or deltoid muscle.
  Safety data were pooled in two comparison groups (Risperidone ISM 75 mg and Risperidone ISM 100 mg) because the sample size increased and therefore the precision around the estimates.
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg
All-Cause Mortality (participants affected / at risk) | 1/116 | 0/99
Serious Adverse Events (participants affected / at risk) | 6/116 | 5/99
Other Adverse Events (participants affected / at risk) | 81/116 | 59/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone ISM 75 mg (N=116) | Risperidone ISM 100 mg (N=99)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 3 (4) | 4 (4)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone ISM 75 mg (N=116) | Risperidone ISM 100 mg (N=99)
Hyperprolactinaemia (Endocrine disorders) | 11 (13) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (2)
Toothache (Gastrointestinal disorders) | 4 (8) | 3 (3)
Asthenia (General disorders) | 7 (8) | 4 (5)
Nasopharyngitis (Infections and infestations) | 13 (15) | 9 (9)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (4)
Weight increased (Investigations) | 8 (9) | 4 (4)
Akathisia (Nervous system disorders) | 4 (4) | 4 (5)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 24 (46) | 18 (29)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4)
Insomnia (Psychiatric disorders) | 13 (16) | 3 (6)
Schizophrenia (Psychiatric disorders) | 5 (9) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor does not object to publication by the Institution of the results of the Trial based on information collected/generated by the Institution. The Institution will provide Sponsor an opportunity to review any proposed publication before it is submitted. If the Trial is part of a multi-center trial, the Institution agress that the first publication is to be a joint publication involving all Trials sites.

DOCUMENTS (3):
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT03870880/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT03870880/SAP_001.pdf
  • Informed Consent Form (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT03870880/ICF_002.pdf